CLINICAL TRIAL: NCT02688686
Title: Safety and Efficacy of DC Vaccine Combined With Cytokine-induced Killer Cells in Patients With Advanced Non-Small-Cell Lung Cancer With Bone Metastases: a Phase I/II Study
Brief Title: Safety and Efficacy of DC-CIK in Patients With Advanced Non-Small-Cell Lung Cancer With Bone Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-CTC-DC/CIK-NSCLC-001
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Non-Small-Cell Lung Cancer With Bone Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: genetically modified dendritic cells + cytokine-induced killer — This Phase I/II Study to evaluate clinical efficacy, safety of genetically modified dendritic cells in combination with cytokine-induced killer cell treament in NSCLC with bone metastases.

SUMMARY:
The purpose of this Phase I/II study is to evaluate the safety and efficacy of dendritic cells(DC) vaccine combined with cytokine-induced killer (CIK) cells in patients with Advanced Non-Small-Cell Lung Cancer with bone metastases. Experimental DC was transfected Ad5 vector coding mRNAs including suppressor of cytokine signaling (SOCS) 1, MUC1 and Survivin,are used for DC-based immunotherapy. Based on the results of our previously preclinical study with DC vaccine combined with CIK cells, the investigators plan to perform the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of non-small cell lung cancer
* Age >18 years at time of consent
* Received standardized treatment of Non-Small-Cell Lung Cancer with bone metastases
* KPS (Karnofsky performance scale) >60
* Patient's written informed consent
* No severe viral or bacterial infections
* Predicted survival >3 months

Exclusion Criteria:

* Clinically relevant diseases or infections (HBV, HCV, HIV)
* Females who are pregnant or nursing
* Immunosuppressant treatment
* Currently participating in another clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
objective response rate (CR+PR) as measured by RECIST criteria | one month after DC/CIK treatment

SECONDARY OUTCOMES:
number of participants with adverse events | 3 days during DC/CIK treatment]

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided